CLINICAL TRIAL: NCT00517426
Title: Effects of Acetazolamide and CO2 Inhalation on Exercise-induced Periodic Breathing in Heart Failure
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Centro Cardiologico Monzino (Other)
Responsible Party: Principal Investigator, Piergiuseppe Agostoni, MD PhD, Centro Cardiologico Monzino
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: R77-CCM S79/407
Record Dates: First submitted 2007-08-16; First posted 2007-08-17 (Estimated); Last update posted 2016-01-28 (Estimated); Status verified 2016-01

CONDITIONS: Chronic Heart Failure
Keywords: heart failure,; exercise; periodic breathing,; acetazolamide
MeSH Terms: conditions — Heart Failure; Motor Activity | interventions — Acetazolamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Active Acetazolamide (Experimental)
  Interventions: Drug: acetazolamide

INTERVENTIONS:
Drug: acetazolamide — i.v. 500 mg of acetazolamide for the acute study and 500 mg of acetazolamide p.o. t.i.d. for two days
  Other Names: Diamox

SUMMARY:
To evaluate the effects of CO2 inhalation and acetazolamide treatment on exercise-induced periodic breathing in patients with chronic stable heart failure.

Patients will be given CO2 (2%) during a constant workload exercise. Patients will be also evaluated by maximal cardiopulmonary exercise test without and with acetazolamide acute and chronic treatment.

ELIGIBILITY:
Inclusion Criteria:

* chronic heart failure in stable clinical condition
* exercise-induced periodic breathing

Exclusion Criteria:

* comorbidities
* NYHA class IV

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2007-07; Primary Completion 2011-07 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Suppression of periodic breathing | two days

SECONDARY OUTCOMES:
suppression of sleeping apnea | two days

CONTACTS AND LOCATIONS:
Overall Officials: Piergiuseppe Agostoni, MD, PhD, Principal Investigator — Centro Cardiologico Monzino
Locations (1):
- Centro Cardiologico Monzino, University of Milan, Milan, Italy

REFERENCES:
- [Background] Agostoni P, Bussotti M, Cattadori G, Margutti E, Contini M, Muratori M, Marenzi G, Fiorentini C. Gas diffusion and alveolar-capillary unit in chronic heart failure. Eur Heart J. 2006 Nov;27(21):2538-43. doi: 10.1093/eurheartj/ehl302. Epub 2006 Oct 6. PMID 17028107